CLINICAL TRIAL: NCT06849284
Title: Idylla™ ThyroidPrint® RUO Assay Beta-Trial Study
Brief Title: To Perform a Post-market Study of the Performance of the Idylla ThyroidPrint Assay Using Clinical Samples in Predicting the Nature of Indeterminate Thyroid Nodules (ITNs) Across Multiple Centers.
Status: Recruiting | Type: Observational
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2425.RCHT.12
Record Dates: First submitted 2024-12-18; First posted 2025-02-27 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To perform a post-market study of the performance of the Idylla™ ThyroidPrint® Assay using clinical samples in predicting the nature of indeterminate thyroid nodules (ITNs) across multiple centers.

DETAILED DESCRIPTION:
This is a multicenter, non-interventional (observational), prospective, post-market study, matching the Idylla™ ThyroidPrint® RUO Assay result to the gold standard of surgical pathology.

The study population is defined as cases where the thyroid nodule has been reported as indeterminate.

Primary endpoints are the calculation of the sensitivity, specificity, and the negative and positive predictive values of the Idylla™ ThyroidPrint® RUO Assay for indeterminate thyroid nodules.

Secondary endpoint: to assess the failure rate of Idylla™ ThyroidPrint® RUO Assay, including errors and invalids; describe the nature of false negative and false positive cases.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid nodule ≥1.0 cm
* With indeterminate cytology
* Surgery due to be performed

Exclusion Criteria:

* Specimens which fail to meet the inclusion criteria.
* FNA fixed in formalin or transferred in alcohol-based collection buffers which is not according to the protocol instructions.
* RNA extracts.
* Patients with ultrasound evidence of malignant cervical adenopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is defined as cases where the thyroid nodule has been reported as indeterminate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary endpoints | Samples taken at Baseline
  to measure the accuracy of the Thyroid print test against the surgical pathology report.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Cornwall Hospital, Truro, Cornwall, United Kingdom